CLINICAL TRIAL: NCT00283478
Title: Randomized Pilot Study of Supplemental Iscar in Combination With Gemcitabine vs. Gemcitabine Alone as Second Line Treatment for Advanced Non-Small Cell Lung Cancer.
Brief Title: Iscar for Second Line Treatment of Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kentuckiana Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1056757; Mistletoe
Record Dates: First submitted 2006-01-26; First posted 2006-01-30 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Advanced stage; Lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Gemcitabine

INTERVENTIONS:
Drug: Iscar Quercus
Drug: Gemcitabine

SUMMARY:
To determine if Iscar Quercus improves immune function and quality of life among patients with stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
RAndomized pilot study of supplemental Iscar in combination with Gemcitabine vs. Gemcitabine alone as second line treatment for advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed IIIB and IV NSCLC who have failed one prior line of chemo
* Karnofsky score 60% or greater
* patients who will be treated with Gemcitabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-05; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To determine if Iscar improves immune function and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Renato V. LaRocca, MD, Study Director — Kentuckiana Cancer Institute
Locations (1):
- Kentuckiana Cancer Institute, Louisville, Kentucky, United States